CLINICAL TRIAL: NCT07042451
Title: Digital Aftercare Assessed: An Evaluation of the Pink Cloud Application in Post-Treatment Substance Use Disorder Support
Brief Title: An Evaluation of the Pink Cloud Application in Post- Treatment Substance Use Disorder Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola Marymount University (Other)
Responsible Party: Principal Investigator, Dr. Joseph LaBrie, Principal Investigator, Loyola Marymount University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R44DA061662 (NIH)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pink Cloud (Experimental): Participants in this arm will receive access to a mobile application designed to support ongoing recovery from substance and alcohol use disorders. The app includes tools that promote engagement with 12-Step recovery principles and offer self-monitoring features. Participants can integrate the app into their recovery efforts as they see fit throughout the study period.
  Interventions: Behavioral: Pink Cloud
- Active Control (Active Comparator): Participants in this arm will receive access to a website containing curated recovery-related materials. These resources are intended to offer general support for individuals in recovery, without emphasizing any specific program or approach. Participants are free to explore and use the content as they choose.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Pink Cloud — Participants randomized to the Pink Cloud condition will receive a subscription code to access the Pink Cloud mobile application for approximately 365 days. The app includes features such as a searchable database of over 245,000 12-Step meetings (in-person and virtual), a sobriety counter, customizable daily planners, personal inventory tools, and a resentment journal. Participants are encouraged to use the app as they see fit throughout the study period. No prompts or required usage schedules will be imposed; instead, engagement will be self-directed to reflect real-world usage patterns.
  Arms: Pink Cloud
Behavioral: Active Control — Participants randomized to the control condition will receive a code to access recovery-related resources hosted on a private study website. These materials include links to mutual-help groups, crisis support services, and educational content and treatment options. Participants may access the website at their discretion and engage with the resources as often and in whatever ways they choose. No prompts or required usage schedules will be imposed.
  Arms: Active Control

SUMMARY:
This randomized controlled trial (RCT) will evaluate the feasibility and efficacy of Pink Cloud, a mobile health application designed to support recovery from substance and alcohol use disorders (SUD/AUD). The app provides access to over 245,000 in-person and virtual 12-Step meetings, along with features such as a sobriety counter, daily planner, and personal inventory tools. In this study, 1,410 participants in various stages of recovery will be randomly assigned to receive either access to the Pink Cloud app or to a control condition. Participants will complete follow-up assessments at 1, 3, and 6 months. Primary outcomes include number of days sober and frequency of drug and alcohol problems. Secondary outcomes include meeting attendance, proportion of sober individuals in one's social network, and engagement in recovery-related activities. The investigators hypothesize that participants in the Pink Cloud group will report more days sober and fewer substance use problems than those in the control group, and that they will also report attending more meetings, having a greater proportion of sober peers, and engaging more frequently in recovery activities.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age or older
* Participant is willing to attend a 12-Step or peer-to-peer recovery meeting (in person or virtual) within the next week
* Participant owns a personal smartphone with cellular service
* Participant is a permanent resident of the United States
* Participant feels comfortable reading and understanding written English in everyday situations
* Participant has consumed alcohol and/or used drugs (excluding tobacco or prescribed medication) at some point in their life, but not within the past couple of days
* Participant is not currently attending outpatient or residential treatment for substance and/or alcohol use
* Participant does not have a plan to enter substance and/or alcohol treatment in the next 30 days
* Participant has been invited by the research team to either the intervention or control condition and redeemed their subscription code.
* Informed consent is provided

Exclusion Criteria:

* Participant is younger than 18 years of age
* Participant is unwilling to attend a 12-Step or peer-to-peer recovery meeting (in person or virtual) within the next week
* Participant does not own a personal smartphone with cellular service
* Participant is not a permanent resident of the United States
* Participant does not feel comfortable reading and understanding written English in everyday situations
* Participant has consumed alcohol or used drugs (excluding tobacco or prescribed medication) within the past couple of days
* Participant has never consumed alcohol or used drugs
* Participant is currently attending outpatient or residential treatment for substance and/or alcohol use
* Participant has a plan to enter substance and/or alcohol treatment in the next 30 days
* Participant was not invited by the research team or did not redeem their assigned subscription code
* Informed consent is not provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1410 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in sobriety status between baseline and 1 month | baseline, 1 month
  Self-reported number of days participant reports not using alcohol or drugs in the past 30 days.
Change in sobriety status between baseline and 3 months | baseline, 3 months
  Self-reported number of days participant reports not using alcohol or drugs in the past 90 days.
Change in sobriety status between baseline and 6 months | baseline, 6 months
  Self-reported number of days participant reports not using alcohol or drugs in the past 180 days.
Change in alcohol and drug problems between baseline and 1 month | baseline, 1 month
  Self-reported frequency of alcohol and drugs problems in the past 30 days.
Change in alcohol and drug problems between baseline and 3 months | baseline, 3 months
  Self-reported frequency of alcohol and drugs problems in the past 90 days.
Change in alcohol and drug problems between baseline and 6 months | baseline, 6 months
  Self-reported frequency of alcohol and drugs problems in the past 180 days.

SECONDARY OUTCOMES:
Change in meeting attendance between baseline and 1 month | baseline, 1 month
  Frequency of 12-Step / peer-to-peer meetings attended in the past 30 days.
Change in meeting attendance between baseline and 3 months | baseline, 3 months
  Frequency of 12-Step / peer-to-peer meetings attended in the past 90 days.
Change in meeting attendance between baseline and 6 months | baseline, 6 months
  Frequency of 12-Step / peer-to-peer meetings attended in the past 180 days.
Change in social network between baseline and 1 month | baseline, 1 month
  Proportion of social network that is sober in the past 30 days.
Change in social network between baseline and 3 months | baseline, 3 months
  Proportion of social network that is sober in the past 90 days.
Change in social network between baseline and 6 months | baseline, 6 months
  Proportion of social network that is sober in the past 180 days.
Change in recovery related activities between baseline and 1 month | baseline, 1 month
  Frequency of engagement with recovery related activities during the past 30 days.
Change in recovery related activities between baseline and 3 months | baseline, 3 months
  Frequency of engagement with recovery related activities during the past 90 days.
Change in recovery related activities between baseline and 6 months | baseline, 6 months
  Frequency of engagement with recovery related activities during the past 180 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola Marymount, Los Angeles, California, United States